CLINICAL TRIAL: NCT03284606
Title: A Pilot Study of the Effect of Taping in the Hemiplegic Patient With a Deficit of the Footbrowers
Brief Title: Effect of Taping in the Hemiplegic Patient With a Deficit of the Footbrowers
Acronym: NEUROTAP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment default
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Groupement Interrégional de Recherche Clinique et d'Innovation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/15/7839; 2016-A01552-49 (Registry Identifier: French ANSM)
Record Dates: First submitted 2017-09-13; First posted 2017-09-15 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAPING (Experimental): taping in conjunction with common rehabilitation for hemiplegic patients
  Interventions: Device: TAPING; Procedure: Common rehabilitation
- NO TAPING (Placebo Comparator): Common rehabilitation for hemiplegic patients without taping
  Interventions: Procedure: Common rehabilitation

INTERVENTIONS:
Device: TAPING — Taping in conjunction with common rehabilitation for hemiplegic patients
  Arms: TAPING
Procedure: Common rehabilitation — Common rehabilitation for hemiplegic patients

SUMMARY:
A majority of people undergoing rehabilitation following a stroke have a deficit of the dorsal flexors of the foot. The implementation of rehabilitation techniques in accordance with the recommendations of learned societies is not sufficient to compensate for this deficit. Also Kinesio Taping's method of Dr. Kenzo Kase has caught our attention by its action on muscle, joint, circulatory and pain functions.

The use of taping would increase the duration of stimulation of the muscles of the dorsiflexors of the foot which would facilitate the motor recovery.

Data from the literature do not support the conclusion that taping is effective, but no studies evaluating the efficacy of this technique in the foot-lift deficiency of the hemiplegic patient have been found.

The investigators hypothesize that the use of taping in conjunction with common rehabilitation for hemiplegic patients following a stroke improves the stimulation of the muscles of the dorsiflexors of the foot with a positive impact on the walking.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a stroke occurring in a period ranging from 15 days to a month before inclusion and presenting left or right hemiplegia.
* Voluntary motricity of the dorsal flexors of the foot greater than or equal to 1 on the scale of Held and Pierrot Deseilligny
* Quadriceps voluntary motor skill greater than or equal to 2 on the scale of Held and Pierrot Deseilligny
* Informed consent of the patient.

Exclusion Criteria:

* - Evolutive neurological disease leading to cognitive impairment (Alzheimer's, Parkinson's, Multiple sclerosis ...)
* Pre-stroke neurological sequelae
* Achilles tendon elongation or tendinous transfer surgery.
* Spasticity of the sural triceps greater than 2 on the modified Ashworth scale
* Injection of botulinum toxin
* Patients under guardianship, curatorships or under safeguard of justice.
* Allergy to glue, skin lesions located on the zone of laying of the bands
* Complex Regional Pain Symptom of the Ankle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
voluntary muscularity | Week 10
  voluntary muscularity measured by the quotation of Held and Pierrot Deseilligny

SECONDARY OUTCOMES:
Spasticity score | Week 10
  Ashworth scale modified for spasticity

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie MORIN, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No